CLINICAL TRIAL: NCT01970189
Title: A Multi-centre, Prospective Disease Registry for Adults Diagnosed With Primary Immune Thrombocytopenia (ITP) in International Countries
Brief Title: The International ITP Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South Eastern Sydney Local Health District (Other Government)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: CTBR-017 (TRA114972)
Record Dates: First submitted 2013-09-19; First posted 2013-10-28 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-07

CONDITIONS: Thrombocytopenia
Keywords: Immune Thrombocytopenia; Primary Immune Thrombocytopenia; Purpura, Thrombocytopenic, Idiopathic; Autoimmune Thrombocytopenia; Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia; Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary Immune Thrombocytopaenia: Recently-diagnosed (i.e. < 6 months) primary ITP adult patients (≥ 18 years) characterized by platelet counts less than 100x109/L as defined by the International Working Group.

SUMMARY:
Primary immune thrombocytopenia (ITP) is an uncommon disease characterised by a low platelet count, which may cause the patient to have a higher risk or increased duration of bleeding. Individual hospitals only encounter a small number of ITP patients each year which makes it difficult to study this disease. By creating this disease registry, we will be able to build a more complete picture of ITP, including treatment practices, through collecting information about the condition from patients across several hospitals in several countries. Research of this kind will help future patients by providing doctors with information about ITP, and about how patients have been treated.

DETAILED DESCRIPTION:
This is an observational disease registry database for recently-diagnosed adult patients with primary ITP that aims to understand the natural history of this rare disease and disease management. Participating investigators will prospectively enter real-world patient data on their enrolled patients with a minimum of 2 years follow up.

Data from this registry will be used to generate descriptive statistics on demographics, clinical characteristics including prevalence and incidence of co-morbidities, treatment patterns, and adverse outcomes (resulting from treatment or disease) on ITP patients on an annual basis. The information will be generated at the national or combined-country level. Furthermore, each institution will have an access to its data and may choose to generate descriptive statistics for its specific institution on a more frequent, ad-hoc basis. New research questions or questions addressing a subset of registry patients to take advantage of combined registry data will require a separate protocol and review by independent committees

The focus of this protocol is on adults with primary ITP, however, in future there may be interest to expand the population to explore secondary ITP patients as well. Hence, this registry is built to allow for some optional preliminary information related to secondary ITP to be captured.

Multi-site participation of this registry project will be rolled out in stages, and will be offered to centres with appropriate expertise. Pilot countries included Australia, Korea, Taiwan, Singapore, Malaysia, Japan, Thailand and Turkey and sites will be selected based on their potential research (interest, resources, and expected patient volume). Additional sites may be added in the future from countries in Asia Pacific, Middle East and Latin America. Japan has an independent national ITP registry run by the government, however voluntary participation of interested Japanese investigators in this database will be welcomed, therefore allowing comparison of data between Japanese and non-Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Recently-diagnosed (i.e. < 6 months) primary ITP adults patients (≥ 18 years) characterized by platelet counts less than 100x109/L as defined by the International Working Group1.
2. Able to provide written consent for data to be included in the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults recently-diagnosed with primary ITP will be prospectively enrolled into the registry. In cases where prospective data collection is not possible from initial diagnosis, eg if sites see mainly referred patients, those patients with pre-existing ITP of no longer than 6 months duration since diagnosis will be allowed into the registry, provided they are still prospectively being followed up or under ongoing review / treatment at the participating institution.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Disease progression of ITP | up to 24 months
  This will include response assessment to each treatment modality, incidence and characteristics of bleeding events, bone marrow results (if available), development of refractory ITP and effects of any medical intervention (whether beneficial or detrimental) in the overall severity of the disease, according to definitions described by the ITP International Working Group.

CONTACTS AND LOCATIONS:
Overall Officials: Beng H Chong, Study Chair — SESLHD
Locations (44):
- Australia (10):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - St George Hospital, Sydney, New South Wales
  - Calvary Mater Newcastle, Sydney, New South Wales
  - Concord Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Flinders Medical Centre, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Vincent's Hospital, Melbourne, Victoria
  - The Alfred, Melbourne, Victoria
- Colombia (3):
  - Foscal, Busaramanga
  - Hemato-Oncologos, Colombia
  - Hospital Pablo Tobón Uribe, Colombia
- Mubarak Alkabeer Hospital, Kuwait City, Kuwait
- Malaysia (3):
  - Penang Hospital, George Town
  - Ampang Hospital, Kuala Lumpur
  - Subang Jaya Medical Centre, Kuala Lumpur
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- South Korea (5):
  - ASAN Medical Centre, Seoul
  - Samsung Medical Centre, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Severance Hospital, Seoul
- Taiwan (5):
  - China Medical University Hospital, Dawan
  - Mackay Memorial Hospital, Dawan
  - National Cheng Kung University Hospital, Dawan
  - Taipei Veteran's General Hospital, Taipei
  - Taichung Veteran's General Hospital, Taiwean
- Thailand (5):
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
  - Chulalongkorn University, Thailand
  - Pramongkutlao College of MEdicine, Thailand
- Turkey (Türkiye) (7):
  - Ankara Numune Training and Research Hosptial, Ankara
  - Ankara Oncology Training and Research Hospital, Ankara
  - Ankara University, Ankara
  - Pamukkale University Medical Faculty, Pamukkale
  - Dokuz Eylul University Medical Faculty, Turkey
  - Erciyes University Medical Faculty, Turkey
  - Gaziantep University Medical Faculty, Turkey
- Uruguay (3):
  - CASMU, Uruguay
  - Hospital Britanico, Uruguay
  - Hospital Militar, Uruguay